CLINICAL TRIAL: NCT01280006
Title: Effect of Selective and Nonselective Cyclooxygenase Enzyme Inhibition on Arterial Blood Pressure and Cerebral Blood Flow With Exposure to Intermittent Hypoxia in Humans
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Marc Poulin, Prof Dr., University of Calgary
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: UC-MMHAP-COX-IH-2010001
Record Dates: First submitted 2011-01-18; First posted 2011-01-20 (Estimated); Last update posted 2011-12-05 (Estimated); Status verified 2011-12

CONDITIONS: Obstructive Sleep Apnea; Hypertension; Cardiovascular Diseases; Stroke
Keywords: Obstructive Sleep Apnea; Hypoxia; Sleep; Blood Pressure; Hypertension; Myocardial Infarction; Stroke; Ventilation; Brain; Cerebral Blood Flow; Renal Blood Flow
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension; Cardiovascular Diseases; Stroke; Hypoxia; Myocardial Infarction; Respiratory Aspiration | interventions — Indomethacin; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Intermittent hypoxia — The subjects will receive five days of drug intervention: either non-selective cyclooxygenase (Indomethacin) or selective cyclooxygenase-2 inhibition (Celecoxib) or placebo. On the testing day, the subjects will undergo an acute intermittent hypoxia testing before and six hours of hypoxic chamber exposure mimicking obstructive sleep apnea syndrome.
Drug: Indomethacin — The subjects will receive five days of drug intervention: either non-selective cyclooxygenase (Indomethacin) or selective cyclooxygenase-2 inhibition (Celecoxib) or placebo. Then they will be tested with an exposure of intermittent hypoxia.
  Indomethacin: 50 mg, Oral, three times per day for five days.
  Other Names: Apo-Indomethacin
Drug: Celecoxib — The subjects will receive five days of drug intervention: either non-selective cyclooxygenase (Indomethacin) or selective cyclooxygenase-2 inhibition (Celecoxib) or placebo. Then they will be tested with an exposure of intermittent hypoxia.
  Celecoxib: 200 mg, Oral, two times per day for five days with a visually matching sequential placebo in between of two doses.
  Other Names: Celebrex
Drug: Placebo — The subjects will receive five days of drug intervention: either non-selective cyclooxygenase (Indomethacin) or selective cyclooxygenase-2 inhibition (Celecoxib) or placebo. Then they will be tested with an exposure of intermittent hypoxia.
  Placebo: Oral, three times per day for five days.

SUMMARY:
The study has been designed to assess the effect of cyclooxygenase inhibition on blood pressure, cerebral blood flow, ventilation and renal hemodynamics following chronic intermittent hypoxia exposure.

DETAILED DESCRIPTION:
The study will specifically evaluate:

1. Cardiovascular effect of cyclooxygenase inhibitors on cerebral, vascular, blood pressure and homeostatic responses following chronic intermittent hypoxia exposure.
2. Ventilatory response of cyclooxygenase inhibitors following chronic intermittent hypoxia exposure
3. Evaluate the renal hemodynamic effect of chronic intermittent hypoxia exposure and cyclooxygenase inhibition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects
* 18 - 45 years of age
* Informed written consent

Exclusion Criteria:

* Any history of cardio-respiratory diseases, ongoing medication, smoking, trauma, acute illnesses, collagen vascular diseases, rheumatoid arthritis, osteoarthritis

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Arterial Blood Pressure | Six weeks
  Blood pressure will be monitored during all three protocols.
Cerebral Blood Flow | Six weeks
  The cerebral blood flow will be mesauresed during each testing days of all three protocols.

SECONDARY OUTCOMES:
Ventilatory Response | Six weeks.
  The ventilatory response will be measured during each testing days of all three protocols.
Renal Hemodynamics | Six weeks
  The renal hemodynamics will be measured during each testing days of all three protocols.

CONTACTS AND LOCATIONS:
Overall Officials: Marc J Poulin, PhD, Principal Investigator — University of Calgary
Locations (1):
- The Laboratory of Human Cerebrovascular Physiology, HMRB 209 & HMRB 230, University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Beaudin AE, Pun M, Yang C, Nicholl DD, Steinback CD, Slater DM, Wynne-Edwards KE, Hanly PJ, Ahmed SB, Poulin MJ. Cyclooxygenases 1 and 2 differentially regulate blood pressure and cerebrovascular responses to acute and chronic intermittent hypoxia: implications for sleep apnea. J Am Heart Assoc. 2014 May 9;3(3):e000875. doi: 10.1161/JAHA.114.000875. PMID 24815497